CLINICAL TRIAL: NCT03391908
Title: A Prospective Monocentric Clinical Study for Multiomics and Imaging-based Assessment of the Vulnerable Coronary Plaques and Associated Risk in Patients Who Presented an Acute Coronary Syndrome
Brief Title: Multiomics and Imaging-based Assessment of Vulnerable Coronary Plaques in Acute Coronary Syndromes
Acronym: MultiPlaque
Status: Completed | Type: Observational
Sponsor: Cardio Med Medical Center (Industry)
Responsible Party: Sponsor
Other Study IDs: CM0116-PLI-1
Record Dates: First submitted 2017-12-31; First posted 2018-01-05 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2021-07

CONDITIONS: Coronary Stenosis; Acute Coronary Syndrome; Acute Myocardial Infarction; Atheromatous Plaques; Atherosclerosis; Unstable Angina; Non-ST Elevation Myocardial Infarction
Keywords: vulnerable plaque, ACS, NSTEMI, vulnerable patient
MeSH Terms: conditions — Coronary Stenosis; Acute Coronary Syndrome; Plaque, Atherosclerotic; Atherosclerosis; Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for determination of miRNA fractions associated with coronary plaque vulnerability
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MP - SG 01: Patients with unstable angina type acute coronary syndrome: patients aged at least 18 years, who have signed the informed consent, and present an unstable angina-type acute coronary syndrome with maximum 48h before presentation, defined as the presence of typical angina pain, with duration of more than 5 minute, accompanied by ECG changes.
  Interventions: Diagnostic Test: cardiac imaging tests
- MP - SG 02: Patients with acute myocardial infarction (STEMI or NSTEMI) that occurred 30 days before randomization: patients aged at least 18 years, who have signed the informed consent, and present with acute myocardial infarction (STEMI or NSTEMI) defined as typical changes on the ECG (ST elevation of minimum 1 mm in at least 2 consecutive leads - STEMI; ST-T changes for NSTEMI) accompanied by increased levels of cardiac troponin I or T, or CK-MB of more than 2x the normal reference value of the laboratory.
  Interventions: Diagnostic Test: cardiac imaging tests

INTERVENTIONS:
Diagnostic Test: cardiac imaging tests — Patients will undergo non-invasive Cardiac Computed Tomography for assessment of coronary plaques and myocardial perfusion, and invasive intracoronary imaging tests (coronary angiography, Intravascular ultrasound, optical coherence tomography and FFR). If imaging will reveal existence of a significant coronary plaque, a percutaneous coronary intervention (PCI - stenting) will be performed.

SUMMARY:
The aim of Multiplaque clinical study is to assess the vulnerability degree of the atheromatous plaques, before and after a myocardial infarction (MI), based on multiomics analysis, associated with invasive and non-invasive data. In this study, a multi-parametric model for risk prediction will be developed, for evaluation of the risk that is associated with the vulnerable coronary plaques in patients that have suffered an acute coronary syndrome.

In the study, evaluation of the imaging characteristics of these coronary plaques will be performed with the use of CT, OCT, IVUS and invasive angiography. We will study the correlation between plaque evolution and (1) the degree of vulnerability at baseline, (2) multiomics profile of the patients and (3) clinical evolution during follow-up.

Also, new techniques for evaluation of the functional significance of coronary stenoses will be studied and validated, such as calculation of the fractional flow reserve or determination of shear stress in areas that are localized within the near vicinity of the vulnerable coronary plaques.

DETAILED DESCRIPTION:
This is a prospective cohort monocentric study.

The primary objective of this study is to research the vulnerability degree of ateromatous plaques before and after a myocardial infarction, based on multiomics data, invasive and non-invasive imaging data, in order to characterize the vulnerable coronary plaque and the vulnerable patient, in patients who have suffered an acute coronary syndrome (unstable angina or acute myocardial infarction).

The secondary objectives of the study are:

* Evaluation of factors associated with the risk for reinfarction in patients with vulnerable plaques, according to their imaging characteristics of vulnerability.
* Evaluation of predictive factors for reinfarction in patients with vulnerable plaques, according to the multiomics profile of the patient.
* Determination of the rate of adverse events and MACE rates (Major Adverse Cardiac Events) according to the vulnerability degree of the coronary plaque at the index moment.
* Evaluation of the efficiency of new methodologies for assessing vulnerable plaques: coronary shear stress determination, trans-stenotic contrast gradient, quantification of coronary plaque components through CT, OCT and IVUS.
* Evaluation of the efficiency of non-invasive methodologies for assessment of the hemodynamic significance of coronary stenoses.

Study population: The study lot will be comprised by 100 patients out of which:

* lot 1 (substudy 1) - 50 patients with unstable angina type acute coronary syndrome
* lot 2 (substudy 2) - 50 patients with acute myocardial infarction (STEMI or NSTEMI) that occurred 30 days before randomization.

Study design and procedures:

Substudy 1: Research of vulnerable plaques in patients with ACS - Unstable angina

Baseline- Day 1: The following procedures will be performed at baseline:

* Personal data recording (age, gender, address, contact);
* anamnesis, cardiovascular risk assessment, comorbidities;
* Physical examination
* Laboratory analysis (biochemistry Cell blood count, troponin assay, hsCRP, matrix metalloproteinases, miRNAs, multiomic analysis)
* ECG
* Echocardiography (LVEF, chamber volumes and diameters, transmitral valvular flow, pulmonary artery pressure, 3D analysis of the regional kinetics with speckle tracking and tissue Doppler, evaluation of valvular regurgitation)
* Myocardial perfusion echocardiography
* Cardiac computed tomography
* Perfusion CT
* Coronary Angiography +/- stent implantation for the culprit lesion
* Optical coherence tomography
* Intravascular ultrasound

Follow-up:

* Month 1 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation
* Month 3 - telephone follow-up
* Month 6 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation
* Month 12 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation
* Month 15 - telephone follow-up
* Month 18 - telephone follow-up
* Month 24 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation, Cardiac Computed Tomography, Perfusion CT

Substudy 2: Research of remaining vulnerable plaques in patients who have suffered an acute myocardial infarction (STEMI or NSTEMI), with maximum 30 days before the enrollment. The index event is considered to be the acute myocardial infarction.

Baseline - day 1: The following procedures will be performed at baseline:

* Personal data recording (age, gender, address, contact);
* Anamnesis, cardiovascular risk assessment, comorbidities;
* Physical examination;
* Laboratory analysis (biochemistry, Cell blood count, troponin assay, hsCRP, matrix metalloproteinases, miRNAs, multiomic analysis)
* ECG
* Echocardiography (LVEF, chamber volumes and diameters, transmitral valvular flow, pulmonary artery pressure, 3D analysis of the regional kinetics with speckle tracking and tissue Doppler, evaluation of valvular regurgitation)
* Myocardial perfusion echocardiography
* Cardiac computed tomography
* Perfusion CT
* Coronary Angiography +/- stent implantation for the culprit lesion
* Optical coherence tomography

Follow-up:

* Month 1 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation
* Month 3 - telephone follow-up
* Month 6 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation
* Month 12 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation
* Month 15 - telephone follow-up
* Month 18 - telephone follow-up
* Month 24 - anamnesis, physical examination, ECG, echocardiography, end-point evaluation, Cardiac Computed Tomography, Perfusion CT

ELIGIBILITY:
Inclusion Criteria:

Substudy 1:

* Patients aged at least 18 years
* Patients who have signed the informed consent
* Unstable angina type acute coronary syndrome with maximum 48h before presentation, defined as the presence of typical angina pain, with duration of more than 5 minute, accompanied by ECG changes.

Substudy 2:

* Patients aged at least 18 years
* Patients who have signed the informed consent
* Acute myocardial infarction (STEMI or NSTEMI) defined as typical changes on the ECG (ST elevation of minimum 1 mm in at least 2 consecutive leads - STEMI; ST-T changes for NSTEMI) accompanied by increased levels of cardiac troponin I or T, or CK-MB of more than 2x the normal reference value of the laboratory.

Exclusion Criteria: (for both substudies)

* Known sensibility for the contrast agents
* Women at reproductive age who does not use contraceptive methods
* Pregnant women
* Any malignancy within the last 5 years
* Acute or chronic renal failure
* Any disease or comorbidity that reduces the life expectancy under 2 years
* Non-compliant patients who, in the opinion of the investigators, will not undergo the follow-up process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study lot will be comprised by 100 patients out of which:
  * lot 1 (substudy 1) - 50 patients with unstable angina type acute coronary syndrome
  * lot 2 (substduy 2) - 50 patients with acute myocardial infarction (STEMI or NSTEMI) that occurred 30 days before randomization.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
rate of major clinical endpoints - acute myocardial infarction - occuring in the follow-up period | 2 years
  The rate of infarction (in the group of unstable angina) or re-infarction (in the group with already established myocardial infarction) will be assessed during the 2-year follow-up and correlated with the degree of plaque vulnerability as determined by imaging tests.

SECONDARY OUTCOMES:
Revascularization rate | 2 years
  The need for revascularization of the culprit lesion and of the non-culprit lesions will be assessed during the 2-year follow-up
Rate of progression of the vulnerability degree of the coronary plaques | 1 year
  The vulnerability degree of each coronary lesion will be assessed by Cardiac CT at base-line and at 1-year follow-up, and the progression/regression of the vulnerability degree will be calculated
MACE rates (Major Adverse Cardiovascular Events) | 2 years
  Major adverse cardiac events represented by cardiac death, all-cause death, rehospitalization rate, target vessel revascularization and re-infarction rate

CONTACTS AND LOCATIONS:
Overall Officials: Theodora Benedek, MD,Prof, Principal Investigator — University of Medicine and Pharmacy of Tirgu Mures, CardioMed Medical Center
Locations (1):
- Cardio Med SRL, Târgu Mureş, Mureș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to other researchers from the same research group and to other collaborating groups and can be used for further statistical sub-analysis
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available immediately after completion of the enrolment and will remain available for at least 5 years

REFERENCES:
- [Result] Benedek T, Jako B, Benedek I. Plaque quantification by coronary CT and intravascular ultrasound identifies a low CT density core as a marker of plaque instability in acute coronary syndromes. Int Heart J. 2014;55(1):22-8. doi: 10.1536/ihj.13-213. Epub 2014 Jan 27. PMID 24463925
- [Result] Benedek T, Gyongyosi M, Benedek I. Multislice computed tomographic coronary angiography for quantitative assessment of culprit lesions in acute coronary syndromes. Can J Cardiol. 2013 Mar;29(3):364-71. doi: 10.1016/j.cjca.2012.11.004. Epub 2013 Jan 17. PMID 23333164
- [Result] Benedek I, Bucur O, Benedek T. Intracoronary infusion of mononuclear bone marrow-derived stem cells is associated with a lower plaque burden after four years. J Atheroscler Thromb. 2014;21(3):217-29. doi: 10.5551/jat.19745. Epub 2013 Oct 12. PMID 24126180